CLINICAL TRIAL: NCT04892069
Title: A Retrospective, Single Centre, Non-interventional Study Investigating the Effect of Ryzodeg® (Insulin Degludec/Insulin Aspart) in a Real-world Adult Population With Type 2 Diabetes in Lebanon
Brief Title: Investigating the Effect of Ryzodeg® in Adult Patients With Type 2 Diabetes in Lebanon
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4597; U1111-1235-6983 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-05-13; First posted 2021-05-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ryzodeg®: Participants are patients with Type 2 Diabetes (T2D) treated with Ryzodeg® (Insulin Degludec/Insulin Aspart) in a real-world adult population in Lebanon
  Interventions: Drug: Insulin Degludec/Insulin Aspart

INTERVENTIONS:
Drug: Insulin Degludec/Insulin Aspart — All patients have been treated at the discretion of the treating physician in accordance with the Ryzodeg® label in Lebanon. Decision to initiate treatment with commercially available Ryzodeg® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.

SUMMARY:
The study is investigating Ryzodeg®,a medication prescribed to patients with type 2 diabetes mellitus.The study is being carried out to investigate the effect of Ryzodeg® on the change of glycated haemoglobin levels and other diabetes indicators. Participants participation will not affect their medical care. In this retrospective study, the study doctor will collect data from the participants patient files available at the study site. Participants will need to sign the informed consent form during a single visit. Participants files will be reviewed and data relevant to the study will be extracted, within 26 weeks before and after Ryzodeg® treatment initiation (total of 52 weeks). Chart review for all patients is expected to take approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female, age above or equal to 18 years at the time of signing the informed consent.
* Patients diagnosed with Type 2 Diabetes Mellitus (T2DM).
* Patients who were not achieving optimal glycaemic control and who required intensification of antidiabetic treatment and Ryzodeg was the treatment of choice.
* Available and documented HbA1c value at less or equal to 12 weeks prior to initiation of Ryzodeg® treatment and end of study within the study windows.
* Available and documented follow up time of at least 52 weeks with 26 weeks follow-up prior to and after initiation of Ryzodeg®.
* The decision to initiate treatment with commercially available Ryzodeg® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as signed informed consent.
* Participation in any clinical study of an approved or non-approved investigational medicinal product within 26 weeks before and after initiation of treatment with Ryzodeg®.
* Having been previously treated with Ryzodeg® prior to study start.
* Female who were pregnant or breast-feeding during the study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are patients with Type 2 Diabetes (T2D) treated with Ryzodeg® (Insulin Degludec/Insulin Aspart) in a real-world adult population in Lebanon
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | From baseline (defined as the time of Ryzodeg® initiation (week -12 to week 0)) to end-of-study (week 26 +/- 6 weeks)
  Percent (%) point. For all primary and secondary outcome measures: Baseline values for effect assessment will be collected as close to and prior to Ryzodeg® initiation as possible (week 0) but none of these values may be more than 12 weeks old. For end of study a window of 6 weeks before and after week 26 is used.

SECONDARY OUTCOMES:
HbA1c less than 7% | At end-of-study week 26
  Percentage of patients
HbA1c less than 7% without any severe hypoglycaemic episodes during period 2 (26 weeks after initiation of Ryzodeg®) | At end-of-study week 26
  Percentage of patients
Change in fasting plasma glucose (FPG) | From baseline to end-of-study week 26
  mmol/L
Change in insulin dose (total, basal, prandial) | From baseline to end-of-study week 26
  units/day
Change in body weight | From baseline to end-of-study week 26
  Kilogram (Kg)
Change in the occurrence of severe hypoglycaemic events before and after initiation of treatment | From week -26 to week 26
  Number of patients experiencing severe hypoglycaemic events in period 1 versus period 2.
  Period 1 is defined as 26 weeks prior to initiation of Ryzodeg® and period 2 is defined as 26 weeks after initiation of Ryzodeg®.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beirut, Hamra, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com